CLINICAL TRIAL: NCT00288509
Title: A Phase III, Prospective, Multicenter, Open-label Extension Study to Assess the Longer Term Safety and Efficacy of Repeated Treatment of Dysport® Intramuscular Injection in the Treatment of Cervical Dystonia
Brief Title: Open-label Extension Study of AbobotulinumtoxinA (Dysport®) for the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-47-52120-731; 2005-002429-29 (EudraCT Number)
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport (Experimental): 250-1000 units
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — In this long-term extension study, a dose of 500 units Dysport was administered by intramuscular injection into the clinically indicated neck muscles in a single dosing session in the first treatment cycle. This was the same dose as given in the preceding study NCT00257660 (Y-47-52120-051). Based on individual safety & efficacy, subjects could then receive up to 3 subsequent injections with doses titrated in 250 unit steps, to a minimum of 250 units and a maximum of 1000 units. Retreatment occurred approximately 12-16 weeks after the previous injection, with the exact timing based on clinical need.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The aim of this study is to assess longer term safety and effectiveness of Dysport®.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the Y-47-52120-051 study, who have completed all study visits up to Week 12, or up to Week 4 in the event of an early withdrawal
* Returned to pre-treatment status as judged by the Investigator

Exclusion Criteria:

* Pure anterocollis or pure retrocollis
* Known antibodies to botulinum toxin type A
* Requirement for botulinum toxin injections to site(s) other than the neck and unable to avoid such treatment for the duration of the study
* Known significant underlying swallowing or respiratory abnormality which might be exacerbated by botulinum toxin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- United States (14):
  - Barrow Neurology Clinics at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - USC School of Medicine, Los Angeles, California
  - University of Florida, Dept of Neurology, Gainesville, Florida
  - University of Miami, Dept of Neurology, Miami, Florida
  - Emory University School of Medicine, Wesley Woods Health Center, Atlanta, Georgia
  - University of Iowa, Dept of Neurology, Iowa City, Iowa
  - Wayne State University Medical Center, Southfield, Michigan
  - Albany Medical Center, Albany, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, Neurological Institute, New York, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwest Medical Center, Movement Disorder Clinic, Dallas, Texas
  - Baylor College of Medicine, Parkinson's Disease Center and Movement Disorders Clinic, Houston, Texas
- Russia (4):
  - Scientific Research Institute of Neurology, RAMS, Moscow
  - Clinic "Cecil Plus", Moscow
  - Municipal Multi-Speciality Hospital #2, Saint Petersburg
  - St Petersburg Pavlov State Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Truong D, Brodsky M, Lew M, Brashear A, Jankovic J, Molho E, Orlova O, Timerbaeva S; Global Dysport Cervical Dystonia Study Group. Long-term efficacy and safety of botulinum toxin type A (Dysport) in cervical dystonia. Parkinsonism Relat Disord. 2010 Jun;16(5):316-23. doi: 10.1016/j.parkreldis.2010.03.002. Epub 2010 Mar 31. PMID 20359934
- [Derived] Mordin M, Masaquel C, Abbott C, Copley-Merriman C. Factors affecting the health-related quality of life of patients with cervical dystonia and impact of treatment with abobotulinumtoxinA (Dysport): results from a randomised, double-blind, placebo-controlled study. BMJ Open. 2014 Oct 16;4(10):e005150. doi: 10.1136/bmjopen-2014-005150. PMID 25324317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed study NCT00257660 (Y-47-52120-051)were recruited in 15 centres in US and 4 centres in Russia from February 2006 to January 2008 to participate in this study NCT00288509 (Y-47-52120-731).
Pre-assignment Details: Of the 116 subjects treated in study NCT00257660, 108 subjects enrolled in this extension study NCT00288509 (Y-47-52120-731). Eight subjects completed study NCT00257660 but elected not to enroll in this extension study.
Period: Treatment Cycle 1
Arm/Group | Dysport
Started | 108
Completed | 102
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Treatment stopped according to protocol | 1
Period: Treatment Cycle 2
Arm/Group | Dysport
Started | 100 (2 subjects completed Cycle 1 but withdrew before Cycle 2 due to insufficient clinical response)
Completed | 97
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 2
Period: Treatment Cycle 3
Arm/Group | Dysport
Started | 96 (One subject completed Cycle 2 but withdrew before Cycle 3 due to insufficient clinical response)
Completed | 91
Not Completed | 5
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Treatment stopped according to protocol | 1
Period: Treatment Cycle 4
Arm/Group | Dysport
Started | 88 (3 subjects completed Cycle 3 but withdrew before Cycle 4, treatment stopped according to protocol)
Completed | 80
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 4
Not completed — Treatment stopped according to protocol | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dysport
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 89
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 81
  Russian Federation | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Toronto Western Spasmodic Torticollis Rating Scale Total Score From Baseline
Description: TWSTRS is comprised of three different components which are severity, disability & pain. There is an ordinal scale for each component and the score range for each is the following: for severity from 0 (absence of severity) to 35 (max severity), for disability from 0 (no disability) to 30 (max disability) and for pain from 0 (no pain) to 20 (max pain). TWSTRS total score is the sum of the 3 component scores, with a range from 0 to a maximum of 85. For each treatment cycle, the change in TWSTRS total score is the score at week 4 minus the score at baseline.
Time Frame: Week 4 follow-up visit
Population: The intention to treat population consisted of all 108 subjects who received Dysport.
  Subjects with incomplete TWSTRS scores were not included in the TWSTRS total score analyses.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 108
points on a scale
  Change in TWSTRS total score for Treatment Cycle 1 | -16.21 (11.54)
  Baseline TWSTRS total score for Treatment Cycle 1 | 42.48 (10.23)
  Week 4 TWSTRS total score for Treatment Cycle 1 | 25.81 (12.83)
  Change in TWSTRS total score for Treatment Cycle 2 | -11.40 (10.83)
  Baseline TWSTRS total score for Treatment Cycle 2 | 34.72 (11.12)
  Week 4 TWSTRS total score for Treatment Cycle 2 | 23.40 (12.55)
  Change in TWSTRS total score for Treatment Cycle 3 | -10.84 (13.00)
  Baseline TWSTRS total score for Treatment Cycle 3 | 32.66 (11.68)
  Week 4 TWSTRS total score for Treatment Cycle 3 | 21.84 (12.45)
  Change in TWSTRS total score for Treatment Cycle 4 | -11.27 (11.46)
  Baseline TWSTRS total score for Treatment Cycle 4 | 34.35 (12.81)
  Week 4 TWSTRS total score for Treatment Cycle 4 | 23.07 (12.62)

2. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale Severity Subscale as a Change From Baseline
Description: TWSTRS is comprised of three different components which are severity, disability & pain. There is an ordinal scale for each component and the score range for severity is from 0 (absence of severity) to 35 (max severity). For each treatment cycle, the change in TWSTRS severity subscale is the score at week 4 minus the score at baseline.
Time Frame: Week 4 follow-up visit
Population: The intention to treat population consisted of all 108 subjects who received Dysport.
  All available TWSTRS severity subscale scores have been included in the severity subscale analyses. Subjects excluded from the TWSTRS total score analyses may have their available data included in the TWSTRS severity subscale score analyses.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 108
points on a scale
  Change in TWSTRS severity score for cycle 1 | -7.68 (5.72)
  Baseline TWSTRS severity score for cycle 1 | 19.79 (4.29)
  Week 4 TWSTRS severity score for cycle 1 | 11.90 (5.54)
  Change in TWSTRS severity score for cycle 2 | -5.52 (5.54)
  Baseline TWSTRS severity score for cycle 2 | 16.05 (5.10)
  Week 4 TWSTRS severity score for cycle 2 | 10.54 (5.43)
  Change in TWSTRS severity score for cycle 3 | -5.68 (6.21)
  Baseline TWSTRS severity score for cycle 3 | 15.79 (5.32)
  Week 4 TWSTRS severity score for cycle 3 | 10.23 (5.95)
  Change in TWSTRS severity score for cycle 4 | -5.78 (5.57)
  Baseline TWSTRS severity score for cycle 4 | 16.53 (5.64)
  Week 4 TWSTRS severity score for cycle 4 | 10.96 (5.95)

3. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale Disability Subscale Score as a Change From Baseline
Description: TWSTRS is comprised of three different components which are severity, disability & pain. There is an ordinal scale for each component and the score range for disability is from 0 (no disability) to 30 (max disability). For each treatment cycle, the change in TWSTRS disability subscale is the score at week 4 minus the score at baseline.
Time Frame: Week 4 follow-up visit
Population: The intention to treat population consisted of all 108 subjects who received Dysport.
  All available TWSTRS disability subscale scores have been included in the disability subscale analyses. Subjects excluded from the TWSTRS total score analyses may have their available data included in the TWSTRS disability subscale score analyses.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 108
points on a scale
  Change in TWSTRS disability score for cycle 1 | -4.25 (4.39)
  Baseline TWSTRS disability score for cycle 1 | 12.70 (4.31)
  Week 4 TWSTRS disability score for cycle 1 | 8.51 (5.22)
  Change in TWSTRS disability score for cycle 2 | -2.88 (3.86)
  Baseline TWSTRS disability score for cycle 2 | 10.45 (4.56)
  Week 4 TWSTRS disability score for cycle 2 | 7.63 (4.83)
  Change in TWSTRS disability score for cycle 3 | -2.74 (4.44)
  Baseline TWSTRS disability score for cycle 3 | 9.73 (4.27)
  Week 4 TWSTRS disability score for cycle 3 | 6.97 (4.67)
  Change in TWSTRS disability score for cycle 4 | -2.54 (3.16)
  Baseline TWSTRS disability score for cycle 4 | 10.09 (4.91)
  Week 4 TWSTRS disability score for cycle 4 | 7.46 (5.07)

4. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale Pain Subscale Score as a Change From Baseline
Description: TWSTRS is comprised of three different components which are severity, disability & pain. There is an ordinal scale for each component and the score range for pain is from 0 (no pain) to 20 (max pain). For each treatment cycle, the change in TWSTRS pain subscale is the score at week 4 minus the score at baseline.
Time Frame: Week 4 follow-up visit
Population: The intention to treat population consisted of all 108 subjects who received Dysport.
  All available TWSTRS pain subscale scores have been included in the pain subscale analyses. Subjects excluded from the TWSTRS total score analyses may have their available data included in the TWSTRS pain subscale score analyses.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 108
points on a scale
  Change in TWSTRS pain score for cycle 1 | -4.53 (4.57)
  Baseline TWSTRS pain score for cycle 1 | 10.08 (4.64)
  Week 4 TWSTRS pain score for cycle 1 | 5.37 (4.97)
  Change in TWSTRS pain score for cycle 2 | -2.99 (4.27)
  Baseline TWSTRS pain score for cycle 2 | 8.12 (5.35)
  Week 4 TWSTRS pain score for cycle 2 | 5.22 (5.34)
  Change in TWSTRS pain score for cycle 3 | -2.41 (5.04)
  Baseline TWSTRS pain score for cycle 3 | 7.16 (5.19)
  Week 4 TWSTRS pain score for cycle 3 | 4.65 (5.01)
  Change in TWSTRS pain score for cycle 4 | -2.81 (4.85)
  Baseline TWSTRS pain score for cycle 4 | 7.72 (5.57)
  Week 4 TWSTRS pain score for cycle 4 | 4.97 (5.14)

ADVERSE EVENTS:
Arm/Group | Dysport
Serious Adverse Events (participants affected / at risk) | 2/108
Other Adverse Events (participants affected / at risk) | 84/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=108)
Appendicitis (Infections and infestations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=108)
Dysphagia (Gastrointestinal disorders) | 27 (45)
Headache (Nervous system disorders) | 7 (8)
Influenza (Infections and infestations) | 10 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 (29)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (13)
Urinary tract infection (Infections and infestations) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication of results from all sites in this multicenter study is expected. If the sponsor no longer plans this or 6 months after study completion at all sites, the PI may publish the results. He will supply any proposed publication to the sponsor for review and comment at least 30 days before submission for publication. If the sponsor believes a patent application should be filed, the publication will be delayed for another 60 days or until patent filing; with a maximum delay of 90 days.